CLINICAL TRIAL: NCT05225571
Title: The Relationship of Cervical Sagittal Parameters With Pain and Disability in Cervical Myofascial Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2021.05.146
Record Dates: First submitted 2021-12-24; First posted 2022-02-04 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Myofascial Pain Syndrome; Neck Pain; Neck Disorder
Keywords: sagittal alignment; myofascial pain syndrome; neck disability; pain intensity
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cervical myofascial pain syndrome: The participants who diagnosed as cervical myofascial pain syndrome aged 18-64 years. The pain must last at least 3 months.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there is no any intervention in this study. it is an observational and cross-sectional study.

SUMMARY:
Participants between the ages of 18-64 who were diagnosed with cervical myofascial pain syndrome will be included in the study. cervical sagittal parameters, numerical pain rating scale, Bournemouth neck questionnaire and cervical range of motion will be measured and evaluated.

DETAILED DESCRIPTION:
It is an observational, cross-sectional study. Participants between the ages of 18-64 who were diagnosed with cervical myofascial pain syndrome, who applied to the Physical Medicine and Rehabilitation Clinic of Kanuni Sultan Süleyman Training and Research Hospital with neck pain for more than 3 months will be included. The pain level of the participants will be evaluated with the numerical pain rating scale, the cervical range of motion and the disability level with the Bournemouth neck questionnaire. C0-2 cervical lordosis angle, C2-C7 cervical lordosis angle, cervical sagittal vertical axis (cSVA), T1 slop, T1 slop - cervical lordosis angle (TS-CL), cervical tilt, thoracic inlet angle (TIA) and Cranial tilt measurement will be performed by using Surgimap software program. The relationship between the level of pain and disability, and cervical sagittal parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age at 18-64 years
* Neck pain due to myofascial pain syndrome for more than 3 months
* Presence of lateral cervical radiograph taken in neutral position in the last 3 months
* Visible lower border of T1 vertebra on lateral radiographs
* Absence of other spinal pathologies such as underlying scoliosis, cervical disc herniation, spondylolysis, spondylolisthesis

Exclusion Criteria:

* Presence of an organic pathology that will cause neck pain
* Inability to see the lower border of the T1 vertebra on lateral cervical radiographs and the radiographs not taken in neutral position

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: The participants who aged 18-64 Years , and diagnosed as cervical myofascial pain syndrome.
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
NRS (Numerical rating scale) | 1 day
  The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which the child rates the pain from 0 (no pain) to 10 (worst pain)
cervical range of motion (degree) | 1 day
  cervical flexion, extension, lateral flexion and rotation angles are actively evaluated.
Bournemouth Neck Questionnaire | 1 day
  Adapted from the Bournemouth Low Back Pain questionnaire developed by Bolton and Humphreys in 2002. The Bournemouth Neck Pain Questionnaire consists of 7 questions in total. Each question scores between 0 and 10. Although the highest score is 70, a high score indicates a high level of disability.
cervical sagittal parameters | 1 day
  Parameters to be checked in cervical lateral radiograph; C0-2 and C2-7 lordosis, T1 slope, c2-7 sagittal vertical axis, TS-CL, servical tilt and cranial tilt.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Damla Korkmaz, Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman TRH, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided